CLINICAL TRIAL: NCT00925145
Title: Single Incision Laparoscopic Appendectomy in the Community Utilizing Conventional Instruments
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Nam Nguyen, University of British Columbia
Other Study IDs: H09-00937
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: Single Incision Laparoscopic Appendectomy

INTERVENTIONS:
Procedure: Single Incision Laparoscopic Appendectomy

SUMMARY:
There is a move to "scarless surgery" and this achieved by doing laparoscopic abdominal surgery though a single small umbilical incision. A technique for laparoscopic appendectomy done through a single incision utilizing conventional instruments has been developed. The operative risk of the single incision approach is no different that the standard three incision laparoscopic appendectomy. The goal is to study the operative time, length of hospital stay, and complications from this operation.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing appendectomy for acute appendicitis

Exclusion Criteria:

* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to a community hospital (RGH) with a working diagnosis of acute appendicitis when the investigator (myself) and co-investigator (Dr. Bloom) are on call for general surgery emergencies.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nam Nguyen, MD, Principal Investigator — University of British Columbia; Scott Bloom, Study Director — University of British Columbia; Connie Chiu, Study Director — University of British Columbia
Locations (1):
- The Richmond Hospital, Richmond, British Columbia, Canada